CLINICAL TRIAL: NCT07298850
Title: A Study on the Effect of CGM Alone on Glycemic Metrics in Type 2 Diabetes Patients Not Using Insulin, Without Additional Interventions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Collaborators: i-SENS, Inc. (Industry)
Responsible Party: Principal Investigator, Sun Joon, Moon, Assistant Professor, Kangbuk Samsung Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KBSMC 2024-06-042
Record Dates: First submitted 2025-12-05; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Continuous Glucose Monitoring; Type 2 Diabetes
Keywords: Type 2 diabetes; Continuous glucose monitoring; Non-insulin Treated Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Sequential CGM Application (Blinded followed by Unblinded) (Experimental): Single arm consisting of adults with non-insulin-treated type 2 diabetes. All participants undergo a 2-week prospective observation using a real-time CGM device (CareSens Air), transitioning from a blinded baseline period to an unblinded intervention period to evaluate glycemic changes.
  Interventions: Device: Continuous glucose monitoring

INTERVENTIONS:
Device: Continuous glucose monitoring — All participants are adults with non-insulin-treated type 2 diabetes. Participants will wear a real-time continuous glucose monitoring (rt-CGM) device (CareSens Air) for a total of two weeks. The intervention consists of two consecutive phases:
  1. Week 1 (Blinded Mode): Participants wear the CGM but cannot view their glucose readings. This period establishes baseline glycemic data.
  2. Week 2 (Unblinded Mode): The same CGM session continues, but the mode is switched to "unblinded." Participants can view their real-time glucose levels and trend arrows.
  Throughout the study, no additional structured education (e.g., diet or exercise coaching) or medication adjustments by the investigators are provided. The study evaluates the effect of data visibility alone on glycemic metrics.

SUMMARY:
This study evaluates the effect of using a real-time continuous glucose monitoring (CGM) system on blood sugar control in people with type 2 diabetes who do not use insulin.

Participants will wear a CGM device (CareSens Air) for a total of two weeks. During the first week, the device will be set to "blinded mode," meaning participants cannot see their glucose readings. During the second week, the device will be switched to "unblinded mode," allowing participants to view their glucose levels and trends in real-time.

The study aims to determine if simply seeing real-time glucose data can help patients improve their blood sugar control (such as increasing the time their blood sugar is in the target range) without receiving additional structured education on diet or exercise. Researchers will compare the glucose data collected during the blinded week with the data from the unblinded week.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Type 2 Diabetes Mellitus (HbA1c ≥ 6.5%, fasting plasma glucose ≥ 126 mg/dL, 2-hour plasma glucose ≥ 200 mg/dL during 75g OGTT, or random plasma glucose ≥ 200 mg/dL with classic symptoms)
2. No medication changes in the past 3 months, and receiving treatment with lifestyle modification or oral antidiabetic drugs or GLP-1 receptor agonists
3. Ages 19 - 80 years old
4. Patients who have voluntarily signed the informed consent form

Exclusion Criteria:

1. Type 1 diabetes patients
2. Insulin users
3. Patients who have changed oral hypoglycemic agents within the past 3 months
4. Patients scheduled for hospitalization within 2 weeks
5. Pregnant women or those planning pregnancy within 1 month
6. Those who do not agree to the program
7. Those deemed unsuitable for participation in this clinical trial by the investigator

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Percentage of Time in Range (TIR) 70-180 mg/dL From Week 1 (Blinded) to Week 2 (Unblinded) | Week 1 and Week 2
  Percentage of time glucose readings are within the target range of 70-180 mg/dL.

SECONDARY OUTCOMES:
Change in Percentage of Time in Tight Range (TITR) 70-140 mg/dL From Week 1 (Blinded) to Week 2 (Unblinded) | Week 1 and Week 2
  Percentage of time glucose readings are within the tight target range of 70-140 mg/dL.
Change in Percentage of Time Below Range (TBR) <70 mg/dL From Week 1 (Blinded) to Week 2 (Unblinded) | Week 1 and Week 2
  Percentage of time glucose readings are below 70 mg/dL, indicating hypoglycemia.
Change in Percentage of Time Below Range (TBR) <54 mg/dL From Week 1 (Blinded) to Week 2 (Unblinded) | Week 1 and Week 2
  Percentage of time glucose readings are below 54 mg/dL, indicating clinically significant hypoglycemia.
Change in Percentage of Time Above Range (TAR) >140 mg/dL From Week 1 (Blinded) to Week 2 (Unblinded) | Week 1 and Week 2
  Percentage of time glucose readings are above 140 mg/dL. This metric assesses exposure to hyperglycemia, including mild elevations.
Change in Percentage of Time Above Range (TAR) >180 mg/dL From Week 1 (Blinded) to Week 2 (Unblinded) | Week 1 and Week 2
  Percentage of time glucose readings are above 180 mg/dL, indicating hyperglycemia.
Change in Percentage of Time Above Range (TAR) >250 mg/dL From Week 1 (Blinded) to Week 2 (Unblinded) | Week 1 and Week 2
  Percentage of time glucose readings are above 250 mg/dL, indicating severe hyperglycemia.
Change in Mean Glucose Concentration From Week 1 (Blinded) to Week 2 (Unblinded) | Week 1 and Week 2
  Average glucose concentration (mg/dL) measured by the CGM device.
Change in Glucose Standard Deviation (SD) From Week 1 (Blinded) to Week 2 (Unblinded) | Week 1 and Week 2
  Standard Deviation (SD) of glucose readings, measuring glycemic variability.
Change in Glucose Coefficient of Variation (CV) From Week 1 (Blinded) to Week 2 (Unblinded) | Week 1 and Week 2
  Coefficient of Variation (CV) calculated as (SD / Mean Glucose) * 100, measuring glycemic variability.
Change in Glucose Management Indicator (GMI) From Week 1 (Blinded) to Week 2 (Unblinded) | Week 1 and Week 2
  GMI is an estimated HbA1c level calculated from the mean glucose concentration derived from CGM data.

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk Samsung Hospital, Seoul, Jongro-Ku, South Korea

IPD SHARING:
Plan to Share IPD: No